CLINICAL TRIAL: NCT00441675
Title: A Long Term Follow up Study for a Comparison of Stepwise Treatment of Asthmatic Children With Salmeterol/Fluticasone Propionate Combination Product (SERETIDE®) and/or Fluticasone Propionate (FLIXOTIDE (TM)) Based on PD20 Methacholine and Symptoms or Based on Symptoms Only.
Brief Title: A Long Term Prospective Follow Up Study For The CATO Study (SAS30018/SER9702)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: SAS107541
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: Adolescents; Asthma; long-term follow-up; symptoms; bronchial hyperresponsiveness
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity

STUDY DESIGN:
Observational Model: Case-Only

GROUPS / COHORTS (2):
- Salmeterol/Fluticasone: Previous Salmeterol/Fluticasone treatment
  Interventions: Procedure: Symptom Score; Procedure: Symptom Score and PD20
- Fluticasone: Previous Fluticasone propionate treatment
  Interventions: Procedure: Symptom Score; Procedure: Symptom Score and PD20

INTERVENTIONS:
Procedure: Symptom Score — Symptom Score
Procedure: Symptom Score and PD20 — Symptom Score and PD20

SUMMARY:
The CATO population is a very well documented population during two years. During this study patients were treated according to the CATO algorithm, after that patient were treated according to the Dutch national (GINA derived) guidelines up to 6 years of follow-up. The purpose of this prospective follow-up study is to understand the long-term effects of treatment. Therefore the measurements done at baseline (CATO part 1) are repeated after 6 years in this CATO-population (CATO follow-up).

DETAILED DESCRIPTION:
A long term follow up study for a comparison of stepwise treatment of asthmatic children with Salmeterol/Fluticasone propionate combination product (Seretide®) and/or Fluticasone propionate (Flixotide®) based on PD20 methacholine and symptoms or based on symptoms only ("Children Asthma Therapy Optimal")

ELIGIBILITY:
Inclusion criteria:

* Any subject who has given informed consent to participate in the CATO study, and has met all the criteria required for randomisation into the clinical study may take part in this follow up study
* Under the age of 18 years Subjects and both parent(s)/guardian(s) who have given written informed consent to participate in the study
* Subjects from 18 years and older who have given written informed consent to participate in the study

Exclusion criteria:

* Experienced an acute asthma exacerbation requiring emergency room treatment within 4 weeks or hospitalisation within 4 weeks of visit 1
* Any use of oral/parenteral or depot corticosteroid within 4 weeks of visit 1
* Subjects who are pregnant (a pregnancy test can be performed at the investigator's discretion)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients randomized in the CATO study (SAS30018) (total of 210) were asked to participate in the follow up study.
  Any subject who gave informed consent to participate in the CATO study, and met all the criteria required for randomisation into the clinical study took part in this follow up study.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the mean annual in FEV1 (% predicted) between randomisation (CATO visit 2) and the current visit 2 between both treatment arms. | 6 years

SECONDARY OUTCOMES:
Comparison of both treatment arms (BHR strategy versus reference strategy):• Lung function FVC and PEFR measured in the clinic between randomisation ( and current visit 2 expressed as the mean annual change of % predicted | 6 years
• Percentage asthma symptom free days during 6 weeks of this extension study • Bronchial hyperresponsiveness, determined with PD20 methacholine between randomisation and current visit 2 | 6 years
Growth rate between randomisation and current visit 2 (expressed as SD-scores)•frequency of asthma exacerbations between randomisation and current visit 2 | 6 years
• Height at current visit 1 or at last measurement at which subject has reached their final height.• Cumulative ICS doses between randomisation and current visit 2 (if this can be achieved with sufficient reliability) | 6 years
Quality of Life (Juniper questionnaire) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Netherlands (14):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Hilversum
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sittard
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Zwolle